CLINICAL TRIAL: NCT07014488
Title: A Single-center, Single-arm, Open-label, Fixed-sequence Study to Evaluate the Effect of Rifampicin on the Pharmacokinetics of Oral HRS-5041 in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of Rifampicin on the Pharmacokinetics of Oral HRS-5041 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-5041-105
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Rifampin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-5041 + Rifampicin (Experimental)
  Interventions: Drug: HRS-5041 Tablets; Drug: Rifampicin Capsule

INTERVENTIONS:
Drug: HRS-5041 Tablets — HRS-5041 tablets.
Drug: Rifampicin Capsule — Rifampicin capsule.

SUMMARY:
The study was designed to evaluate the pharmacokinetic effects of Rifampicin on HRS-5041 after oral administration of HRS-5041 tablets in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged 18-55 years (inclusive).
2. Male participants whose partner was a woman of childbearing potential were required to use contraception from the time they provided written informed consent until 3 months after the last dose of the investigational product.
3. Weight ≥ 50 kg and body mass index (BMI) : 19-28 kg/m2 (inclusive).
4. Participants were able to communicate well with the investigators, understand and comply with the requirements of the study, and sign the informed consent form.

Exclusion Criteria:

1. Patients who have had or are currently suffering from any clinically serious diseases of the circulatory system, endocrine system, nervous system, digestive system, respiratory system, genitourinary system, hematology, immunology, psychiatry or metabolic system or any other diseases that may interfere with the test results.
2. Patients who had undergone surgery within 6 months before screening or who were scheduled to undergo surgery during the study or who had undergone any previous surgery affecting gastrointestinal absorption (including gastrectomy, bowel resection, or gastric contraction).
3. Patients who had donated blood or had massive blood loss (≥400 mL), received blood transfusion, or used blood products within 3 months before screening.
4. Allergic constitution, including severe drug allergy or history of drug allergy; He had a history of allergy to HRS-5041 tablets, rifampicin, or their excipients.
5. History of drug abuse within 1 year before screening; Those with positive urine drug abuse screening.
6. Who participated in any clinical trial and took a study drug within 3 months before the first dose.
7. Drinking more than 14 units of alcohol per week in the 6 months prior to screening (1 unit = 285 mL for beer, 25 mL for spirits, or 100 mL for wine); Or have taken alcohol-containing products 48 hours before administration; Or positive alcohol breath test at baseline.
8. Patients with abnormal vital signs and judged by the investigator to be clinically significant.
9. HCV (hepatitis C virus) antibody positive, HIV antibody positive, HBsAg positive, syphilis antibody positive.
10. Those who have special requirements for diet and cannot abide by the uniform diet.
11. Patients with a history of needle fainting and blood fainting, difficulty in blood collection or inability to tolerate venous puncture blood collection.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-06-20 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve from time 0 to time t (AUC0-t) | 0 to anticipated 23 days.
Area Under the Curve from time 0 to infinity (AUC0-∞) | 0 to anticipated 23 days.
Maximum concentration (Cmax) | 0 to anticipated 23 days.

SECONDARY OUTCOMES:
Time to reach maximum concentration (Tmax) | 0 to anticipated 23 days.
Half-life (t1/2) | 0 to anticipated 23 days.
Apparent clearance (CL/F) | 0 to anticipated 23 days.
Adverse events (AEs) | 0 to anticipated 31 days.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University (Shandong Provincial Qianfoshan Hospital), Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided